CLINICAL TRIAL: NCT00332930
Title: An Extension Study to Protocol VIR-NCHR-01 to Assess the Antiretrovirological Properties of a Therapeutic HIV Vaccine Candidate Based on Recombinant Fowlpox Virus (rFPV) (ITV Extension Study)
Brief Title: ITV Extension Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); Virax Pty. Ltd, (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIR-NCHR-02
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2006-06

CONDITIONS: HIV
Keywords: HIV; Therapeutic vaccine
MeSH Terms: interventions — Interferon-gamma

INTERVENTIONS:
Biological: recombinant fowlpoxvirus (rFPV) expressing HIV gag-pol antigens
Biological: HIV gag-pol antigens and interferon-gamma (IFN-y)

SUMMARY:
The objective of this phase I/II therapeutic human immunodeficiency virus (HIV) vaccine candidate study is to provide proof of concept for a HIV antigen delivery system in terms of safety, virological effects and selected immune responses in HIV infected individuals after cessation of antiretroviral combination therapy (ART).

DETAILED DESCRIPTION:
A multi-centre, double-blind, placebo-controlled, 20-week parallel group extension study to the VIR-NCHR-01 protocol (ITV study). The purpose of the extension study is to assess the safety and virological effects of a therapeutic HIV vaccine strategy in HIV-1 infected adults currently enrolled in the ITV study after cessation of antiretroviral therapy. Two active candidate vaccines will be studied in this trial: The active treatment arms will receive recombinant fowlpoxvirus (rFPV) expressing HIV gag-pol antigens or HIV gag-pol antigens and interferon-gamma (IFN-y) in diluent. Vaccines will be delivered by intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected individuals eligible and still fulfilling the criteria for the VIR-NCHR-01 protocol (ITV study)
* Received all 3 immunisations
* Remained in follow-up for at least 52 weeks
* Continued to take combination antiretroviral therapy with no evidence of treatment failure at the time entering the roll-over phase
* Written informed consent obtained

Criteria for Withdrawal of Study Participants

* Incidental or progression of disease which, in the opinion of the principal investigator, should preclude further study participation
* If the study participant required cytotoxic or immunosuppressive chemo- or radiation therapy
* If the study participant required any medications that when combined with the study vaccination, would in the opinion of the principal investigator, jeopardise the validity of the individual's continued participation
* Administration of prohibited alternative therapy
* Study participant non-compliance
* All study participants are required to adhere to the protocol evaluation schedule. Failure to adhere with this schedule without having first provided justification may result in the participant being withdrawn from the study
* At the request of the study participant or principal investigator without prejudice to future health care
* In the opinion of the investigator, if it is not in the patient's best interests to continue the study
* At the request of the National Centre in HIV Epidemiology and Clinical Research (NCHECR) with reasonable cause
* At the advice of the Data Safety Monitoring Board (DSMB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2002-09; Study Completion 2003-09

PRIMARY OUTCOMES:
Time weighted area under the curve change from plasma HIV-RNA VL at baseline (day 0) until reintroduction of antiretroviral therapy

SECONDARY OUTCOMES:
Log plasma HIV-RNA load after cessation of combination ART (post-vaccination viral load (VL) set-point)
Kinetics and rate of VL recrudescence and median time to re-initiation of ART
CD8+ T-cell responses to HIV antigens assessed through:
Enzyme linked immunospot (ELISPOT) assay of IFN-y secreting cells
Intracellular Cytokine Cytometry (ICC) for IFN-y and CD69
Human Leucocyte Antigen (HLA) class I/ I matched tetramer analyses for HIV epitope specific CD8+/CD4+ T -cells
CD4+/CD8+ T-cell count changes

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, AO DSc MD FRACP FRCPA FRCP, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.
Locations (6):
- Australia (6):
  - 407 Doctors, Sydney, New South Wales
  - Ground Zero Medical Practice, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - St Vincents Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Carlton Clinic, Melbourne, Victoria